CLINICAL TRIAL: NCT03726710
Title: Telemedicine and the Barbershop Model of Hypertension Care for Black Men
Brief Title: Cut Your Blood Pressure 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Medtronic Foundation (Unknown); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Florian Rader, Co-Director, Clinic for Hypertrophic Cardiomyopathy and Aortopathies ; Assistant Director, Non-invasive Laboratory; Hypertension Center of Excellence, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 54480
Record Dates: First submitted 2018-10-30; First posted 2018-10-31 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Hypertension; High Blood Pressure; African American Men
MeSH Terms: conditions — Hypertension | interventions — Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood Pressure measurement and pharmacy (Experimental): Blood Pressure measurement performed by barber and Blood pressure measurement and management visits with study pharmacist in person and through Telemedicine.
  Interventions: Behavioral: Blood Pressure measurement and pharmacy

INTERVENTIONS:
Behavioral: Blood Pressure measurement and pharmacy — Blood Pressure monitoring by barber, Blood pressure measurement and management by pharmacist in person and through telemedicine

SUMMARY:
The recently published LA Barbershop in the New England Journal of Medicine (Victor et al. N Engl J Med 2018; 378: 1291-301) solid evidence of the efficacy of a pharmacist-led medication management intervention to reduce blood pressure in black men that patronize barbershops.

One of the most significant logistical inefficiencies of the LA Barbershop Study was the amount of time the pharmacists spent driving for face-to-face visits with participants. On average, each round trip was 40 miles and pharmacists drove 2 hours per day. By using telemedicine, the study team can minimize the number of face-to-face in-person visits and increase pharmacist efficiency by 25%. the study team aim to increase the scalability of our novel, evidence-based barbershop model by addressing this inefficiency with the pilot study.

In the LA Barbershop trial, each participant averaged 7 in-person visits in 6 months. the study team found that the initial in-person visits between the pharmacist, barber, and patron were essential for establishing trust as well as obtaining baseline electrolyte and serum creatinine levels (with our validated point-of-care device, iSTAT). However, once rapport has been established and blood pressure control achieved, the study team postulate that the effect can be maintained remotely with telemedicine. Our data indicate that most patients' can achieve their blood pressure goal in 3 months or less. the study team propose replacing additional in-person visits with telemonitoring (via Skype or FaceTime) at this juncture, provided blood chemistries are stable.

the study team plan to pilot this in 20 patients from 2 to 3 barbershops for 12 months.

DETAILED DESCRIPTION:
recently published in the New England Journal of Medicine (Victor et al. N Engl J Med 2018; 378: 1291-301) solid evidence of the efficacy of a pharmacist-led medication management intervention to reduce blood pressure in black men that patronize barbershops.

the study enrolled a cohort of 319 hypertensive non-Hispanic black male patrons from 52 black-owned barbershops in Los Angeles County into a cluster-randomized trial in which barbershops (non-traditional health care setting) were assigned to either a pharmacist-led intervention (in which barbers encouraged in-person meetings with pharmacists who then prescribed drug therapy under a collaborative practice agreement with the participants' doctors) or an active control approach (in which barbers encouraged lifestyle modification and doctor appointments).

At 6 months, the mean systolic blood pressure fell by 27.0 mmHg in the intervention group and by 9.3 mmHg in the control group. A blood pressure level of less than 130/80 was achieved in 64% of the participants in the intervention versus 12% of participants in the control group.

the study team are applying for this grant as a first step in transitioning this evidence-based intervention into a scalable program. Specifically, the study team will do a pilotstudy to test whether the impressive effects on blood pressure can be maintained just as well if face-to face meetings are substituted with telemonitoring after blood pressure is at goal. If successful this approach would markedly increase efficiency by increasing the number of patients a single pharmacist can manage.

Non-Hispanic black men have the highest rate of hypertension-related death of any racial, ethnic, or sex group in the United States. Black men have less physician interaction than black women and lower rates of hypertension treatment and control, necessitating community outreach. Because black men with hypertension often have multiple cardiovascular risk factors, marked reductions in blood pressure - if sustained with the use of our approach and then initiated more widely - might reduce the high rates of hypertension-related disability and death among black men in the United States.

The study team want to demonstrate that participants in this pilot can achieve similar blood pressure reduction at 12 months (as compared to those in our previous trial) when telemedicine is substituted for in-person pharmacist visits after 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Non-Hispanic Black Men
* Age 35 to 79 years-old
* Able to give informed consent
* Long-term/frequent barbershop patronage (>8 haircuts at the same barbershop in the last 12 months)
* systolic BP ≥140 on 2 different screening days, and complete set of baseline data
* Each participant should have their own personal smart cell phone with video chat capability (needed for telemedicine)

Exclusion Criteria:

* Women
* Men < 35 years old or Men >79 years old
* Non-black
* Hispanic Ethnicity
* New/infrequent patronage (<8 haircuts at same barbershop in last 12 months);
* Kidney dialysis.
* Receiving chemotherapy for cancer. Systolic BP <140 at either screening and incomplete baseline data.

Ages: 35 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Primary Blood Pressure Outcome - Change in Systolic Blood Pressure | 6 months
  The Pre-Specified primary outcome was the change in systolic blood pressure from baseline to 6 months follow-up.
Primary Blood Pressure Outcome - Change in Systolic Blood Pressure | 12 months
  The Pre-Specified primary outcome was the change in systolic blood pressure from baseline to 12 months follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Blyler CA, Ebinger J, Rashid M, Moy NP, Cheng S, Albert CM, Rader F. Improving Efficiency of the Barbershop Model of Hypertension Care for Black Men With Virtual Visits. J Am Heart Assoc. 2021 Jul 6;10(13):e020796. doi: 10.1161/JAHA.120.020796. Epub 2021 Jun 22. PMID 34155907